CLINICAL TRIAL: NCT03227094
Title: Simplification of CF-related Diabetes Screening by the Use of a Home-based Oral Glucose Tolerance Test (OGTT): A Pilot Study to Evaluate the Validity and Patients' Perceptions
Brief Title: Simplification of CF-related Diabetes Screening at Home
Acronym: AtHome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Université de Montréal (Other); Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: AtHome
Record Dates: First submitted 2017-07-18; First posted 2017-07-24 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis-related Diabetes
Keywords: Diabetes; Screening test; Continuous glucose monitoring; Oral glucose tolerance test
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus | interventions — Beverages; Candy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard OGTT (Other): OGTT standard test at hospital (75g glucose beverage; 2-h test with plasma glucose collection)
  Interventions: Diagnostic Test: Standard OGTT
- Home-based OGTT (Beverage) (Experimental): Home-based OGTT with CGM device, without glucose collection (75g glucose beverage; 2-h test: glycemia measured by CGM)
  Interventions: Diagnostic Test: Home-based OGTT (Beverage)
- Home-based OGTT (Candy) (Experimental): Home-based OGTT with CGM device, without glucose collection (75g of glucose (Jelly Beans); 2-h test: glycemia measured by CGM)
  Interventions: Diagnostic Test: Home-based OGTT (Candy)

INTERVENTIONS:
Diagnostic Test: Standard OGTT — Standard-OGTT Plasma glucose : 0, 30, 60, 90, 120 minutes Complete biochemical profile, weight and size (body mass index), drugs list, pulmonary function by spirometry (FEV, etc.) Questionnaires CGMS training & delivery of Jelly-Bean/75g glucose beverage
  Arms: Standard OGTT
Diagnostic Test: Home-based OGTT (Beverage) — In a random order Candy-OGTT (Jelly-Bean) or 75 g glucose beverage Glycemia every 15 minutes from CGMS collection; standardized condition (fasting + rest) Questionnaires
  Arms: Home-based OGTT (Beverage)
Diagnostic Test: Home-based OGTT (Candy) — In a random order Candy-OGTT (Jelly-Bean) or 75 g glucose beverage Glycemia every 15 minutes from CGMS collection; standardized condition (fasting + rest) Questionnaires
  Arms: Home-based OGTT (Candy)

SUMMARY:
Cystic fibrosis (CF)-related diabetes (CFRD) is the most common complication after pulmonary complications. This specific form of diabetes is associated with an increased morbidity and mortality. CFRD prevalence at the age of 10 is 10% and reaches 40 to 50% in adulthood, while another 35% of adult patients presents impaired glucose tolerance.

In order to identify patients at risk and to implement early therapeutic measures, an annual CFRD screening test should therefore be undertaken for CF patients after 10 years of age. The 2-hour oral glucose tolerance test (OGTT) with a sweet beverage is the recommended screening test. However, participation rates for screening tests are far from optimal. For examples, in 2015, the investigators observed that only 47% of non-diabetic patients attended to planned screening despite large availability and advertisement (unpublished data). Comparable low levels of screening for CFRD, usually below 33%, have been reported by various teams. Several reasons could explain these low adherence rates. Some factors are related to patients perceptions and experience: OGTT is perceived as an additional medical burden requiring a scheduled appointment (several weeks after the last exacerbation); overnight fasting followed by the intake of a large glucose load within 5 minutes can lead to nausea, headache, bloating and fatigue; some patients fear multiple blood sampling, etc. In addition, in case of CFRD diagnosis, recommended capillary blood glucose monitoring, nutritional advice and treatment (insulin) are perceived as extremely invasive and complex, thus some patients prefer avoiding screening test. To date, no alternative screening method has demonstrated its effectiveness to screen for CFRD. The investigators of this study believe that a simplified version of the OGTT would be more attractive, would make it more acceptable for patients and has the potential to improve their adherence to screening tests, simplify CF-team works and reduce costs. By allowing appropriate education and introduction of treatment in a timely manner, improved adherence to annual screening for dysglycemia has the potential to minimize or prevent clinical deterioration observed in years preceding CFRD onset.

DETAILED DESCRIPTION:
The investigators propose a pilot study to evaluate the validity and the acceptability of a home-based OGTT by comparing, in patients with CF:

* Standard hospital-based OGTT with measures of plasma glucose and the use of 75g glucose beverage;
* Home-based OGTT with measures of glucose using a continuous glucose monitoring system (CGMS; without blood sample collection) and the 75g glucose beverage;
* Home-based OGTT with measures of glucose using CGMS and 75g of glucose from candies as a substitute to this poorly appreciate beverage.

Specific objectives are to determine i) the internal validity (specificity, sensitivity) of both home-based OGTTs versus a standard OGTT in controlled setting, and ii) the predictive value (positive and negative). The investigators will also iii) investigate patient's perception and likelihood that the proposed method improves adherence to annual screening, and iv) evaluate potential cost reduction associated with proposed simplified screening tests.

On the day of the OGTT, and after obtaining informed consent, a CGMS will be installed. Patients will receive the very simple training required to use it as well as a pre-packed Jelly Beans bag containing 75g of glucose and a standard 75g glucose beverage bottle. This CGMS will provide interstitial glucose values each 15 min over the next 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult CF-patient without known diabetes
* In stable condition at least 1-month apart from the last exacerbation.

Exclusion Criteria:

* Known CFRD
* Recent exacerbation
* Use medications known to interfere with glucose metabolism such as oral steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Internal validity | OGTTs performed within 14 days
  Specificity and sensitivity of both home-based OGTTs versus a standard OGTT in controlled setting
Predictive value (positive and negative) | OGTTs performed within 14 days
  Both home-based OGTTs versus a standard OGTT in controlled setting

SECONDARY OUTCOMES:
Patient's perception | OGTTs performed within 14 days
  Visual analog scale questionnaire
Cost evaluation of methods | OGTTs performed within 14 days
  Estimated cost of each methods

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Montreal Research Clinical Institute
Locations (2):
- Canada (2):
  - Montreal Clinical Research Institute (IRCM), Montreal, Quebec
  - CHUM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No